CLINICAL TRIAL: NCT01050647
Title: Progesterone for the Management of Preterm, Premature Rupture of the Membranes: A Randomized Controlled Trial.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Professor of Obstetrics and Gynecology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-01082010-4683; 17976 (Other: Stanford University Medical Center)
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 17-hydroxyprogesterone caproate (Active Comparator): Weekly injections of 17-hydroxyprogesterone caproate until patient reached 34 completed weeks of gestation
  Interventions: Drug: 17-Hydroxyprogesterone Caproate
- Castor oil injections (Placebo Comparator): Weekly injections of Caster Oil (placebo)
  Interventions: Other: Caster Oil injections

INTERVENTIONS:
Drug: 17-Hydroxyprogesterone Caproate — Weekly injections of 17-hydroxyprogesterone caproate.
  Other Names: Active study drug
  Arms: 17-hydroxyprogesterone caproate
Other: Caster Oil injections — Weekly injection of Caster Oil (Placebo) until patient reached 34 weeks gestation.
  Other Names: Placebo
  Arms: Castor oil injections

SUMMARY:
Preterm birth is the leading cause of neonatal death and a significant cause of life long disability and health problems. It has been shown that the drug 17-hydroxyprogesterone caproate can help reduce the risk of preterm delivery in women with certain risk factors for preterm birth. We hope to learn whether this same medication can be used to prolong pregnancy in a group of patients in whom this medication has not been previously studied. Specifically, we hope to learn whether progesterone supplementation will delay delivery in women with pre-term, premature rupture of membranes (PPROM).

DETAILED DESCRIPTION:
When women present to either the Obstetrical clinic or labor and delivery with a complaint of possible preterm, premature rupture of membranes (PPROM), they will be examined by an obstetrician to either confirm or rule out this diagnosis. If they are diagnosed with PPROM, they will then be admitted to Lucile Packard Children's Hospital and treated with the normal protocol which includes receiving antibiotics, receiving steroids, being hospitalized until delivery, and having ongoing maternal and fetal monitoring for possible complications. The patients will be identified by their treating obstetricians as possible study candidates and asked by a member of the treatment team if they are potentially interested in participating in a research study. Subsequently, a member of the study team or the treating physician will approach the patient about participating in the trial. Those who choose to participate will receive the standard care protocol in addition to receiving the study medication. The study medication will be a weekly injection of either placebo or 17-hydroxyprogesterone caproate or placebo. The placebo medication (castor oil) was chosen as it has been used in previous studies as a placebo for 17-hydroxyprogesterone caproate. The choice of which medication the patient receives will be determined by a randomization table. Only the pharmacist will be aware of the medication that has been administered. The patient, members of the treatment team, and members of the study team will be blinded to the medication that is being administered. The timing of their delivery will be managed by the treating obstetrician according to standard medical practice. After delivery, the patient's and her infant's medical outcomes will be recorded for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. 18yr of age
2. Singleton pregnancy
3. PPROM confirmed on clinical exam
4. GA between 24+0 and 33+5 wk
5. Ability to understand consent in either English or Spanish

Exclusion Criteria:

1. Contraindication to ongoing pregnancy including:

   1. Evidence of active infection
   2. Evidence of significant placental abruption
   3. IUFD diagnosed at the time of P-PROM diagnosis
2. Major fetal malformation
3. Maternal allergy to progesterone or placebo drug components
4. Current use of progesterone at the time of P-PROM
5. Multiple Gestations
6. Inability to understand consent in either English or Spanish

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Y El-Sayed, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (1.9) | 31.7 (2.0) | 31.7 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21
History of prior preterm birth [Count of Participants; unit: Participants] | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Achievement of 34 Weeks Gestation
Description: Delayed delivery until 34 weeks gestation.
Time Frame: From enrollment until delivery, an average of 34 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Neonatal Respiratory Distress Syndrome
Time Frame: From delivery until neonatal hospital discharge, assessed up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Number analyzed (Participants) | 10 | 11
Participants | 7 | 10
Statistical Analysis 1: Comparison: 17-hydroxyprogesterone Caproate vs Castor Oil Injections; Test type: Superiority; p = 0.31, Chi-squared

3. Secondary Outcome: Number of Participants With Neonatal Grade III - IV Intraventricular Hemorrhage
Time Frame: From delivery until neonatal hospital discharge, assessed up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Number analyzed (Participants) | 10 | 11
Participants | 1 | 2
Statistical Analysis 1: Comparison: 17-hydroxyprogesterone Caproate vs Castor Oil Injections; Test type: Superiority; p > 0.99, Chi-squared

4. Secondary Outcome: Number of Participants With Neonatal Necrotizing Enterocolitis
Time Frame: From delivery to neonatal discharge, assessed up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Number analyzed (Participants) | 10 | 11
Participants | 2 | 1
Statistical Analysis 1: Comparison: 17-hydroxyprogesterone Caproate vs Castor Oil Injections; Test type: Superiority; p = 0.59, Chi-squared

5. Secondary Outcome: Neonatal Length of NICU and Total Hospital Stay Assessed as Number of Days
Time Frame: From birth to discharge form delivery hospital, assessed up to 2 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Number analyzed (Participants) | 10 | 11
days | 39 [13 to 59] | 50 [34 to 69]
Statistical Analysis 1: Comparison: 17-hydroxyprogesterone Caproate vs Castor Oil Injections; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Length of Latency Assessed as Number of Days
Time Frame: From rupture of membranes until delivery, assessed up to 34 weeks of gestation
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
Number analyzed (Participants) | 10 | 11
days | 14.5 [8.9 to 29.1] | 8 [5.3 to 13.4]
Statistical Analysis 1: Comparison: 17-hydroxyprogesterone Caproate vs Castor Oil Injections; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From enrollment up to discharge from the delivery hospital, assessed up to 2 months after delivery
Arm/Group | 17-hydroxyprogesterone Caproate | Castor Oil Injections
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No